CLINICAL TRIAL: NCT06974136
Title: Transcranial Electrical Stimulation Modalities for the Treatment of Clinical Symptoms and Cognitive Deficits in Attention-deficit Hyperactivity Disorder Disorder
Brief Title: tES Modalities for the Treatment of ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Leibniz Research Centre for Working Environment and Human Factors (Other); RWTH Aachen University (Other); Institute for Research in Fundamental Sciences (Unknown)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, The National Brain Mapping Laboratory (NBML)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IPM-NDD
Record Dates: First submitted 2025-04-30; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Neurodevelopmental Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active tDCS group (Active Comparator): This group receives Transcranial Direct Current Stimulation (tDCS). tDCS delivers a constant, low-intensity direct current (typically 1-2 mA) through electrodes placed on the scalp. The anode (positive electrode) increases cortical excitability by depolarizing neurons, while the cathode (negative electrode) decreases excitability by hyperpolarizing neurons.
  Interventions: Device: transcranial electrical stimulation
- active tACS group (Active Comparator): This group receives Transcranial Alternating Current Stimulation (tACS). tACS applies an oscillating current at specific frequencies (e.g., 1-100 Hz) to entrain or synchronize neural oscillations. By aligning the stimulation frequency with endogenous brain rhythms (e.g., theta or gamma bands), tACS can modulate network dynamics, potentially normalizing aberrant oscillatory patterns associated with disorders like ADHD.
  Interventions: Device: transcranial electrical stimulation
- sham group (Placebo Comparator): This group receives sham stimulation. The stimulation duration is for 1 minuetand the device will be turned off after the stimulation
  Interventions: Device: transcranial electrical stimulation

INTERVENTIONS:
Device: transcranial electrical stimulation — Transcranial electrical stimulation (tES) is a non-invasive neuromodulation technique that applies low-intensity electrical currents to the scalp to modulate brain activity. It targets specific brain regions to influence neuronal excitability, connectivity, and plasticity, offering potential therapeutic benefits for neurological and psychiatric conditions. tES is portable, cost-effective, and generally well-tolerated, with minimal side effects such as mild tingling or itching at the stimulation site.
  Other Names: tDCS; tACS

SUMMARY:
This project investigates the efficacy of transcranial electrical stimulation (tES) modalities, specifically transcranial direct current stimulation (tDCS) and transcranial alternating current stimulation (tACS), for treating Attention-Deficit/Hyperactivity Disorder (ADHD) in children and adolescents.

DETAILED DESCRIPTION:
This project aims to evaluate the therapeutic potential of transcranial electrical stimulation (tES) modalities, specifically transcranial direct current stimulation (tDCS) and transcranial alternating current stimulation (tACS), as innovative, non-invasive interventions for managing Attention-Deficit/Hyperactivity Disorder (ADHD) in children and adolescents. ADHD is a neurodevelopmental disorder characterized by persistent inattention, hyperactivity, and impulsivity that impair daily functioning. Conventional treatments, such as pharmacological interventions and behavioral therapies, may have limitations, including side effects or variable efficacy, prompting the exploration of neuromodulation techniques like tES.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD by a licensed psychiatrist and a behavioral checklist
* being 7-18 years old
* providing written informed consent signed by parents

Exclusion Criteria:

* comorbidity with other neurodevelopmental disorders
* Comorbidity with other neurological disorders
* previous history of neurosurgery
* Presence of any ferromagnetic metal in the head
* implanted medical devices in the head or neck region
* history of non-controlled epilepsy with seizures in the last year

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
ADHD symptoms- Clinical rating scale | Baseline, week 2, up to 1 month after the intervention
  ADHD symptoms will be assessed using a DSM-based structured interview. This approach involves a systematic, standardized method to evaluate the presence and severity of ADHD symptoms based on the diagnostic criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders (DSM), likely the DSM-5, which is widely used for diagnosing ADHD.

SECONDARY OUTCOMES:
Executive function- Performance accuracy and reaction time | Baseline, week 2, up to 1 month after the intervention
  Performance in an executive functions computerized task
electroencephalogram (EEG) power | Baseline, week 2
  Change in the EEG alpha/theta/gamma power
electroencephalogram (EEG) functional connectivity | Baseline, week 2

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Research in Fundamental Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided